CLINICAL TRIAL: NCT00919607
Title: Evaluate the Pharmacokinetics of Quetiapine Fumarate in Chinese Schizophrenic Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: D1444C00007
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Last update posted 2010-03-26 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia
Keywords: quetiapine fumarate(SEROQUEL) extended-release(XR) China PK Study; pharmacokinetics parameters
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): quetiapine fumarate extended-release 300mg,administered once-daily Day1~5
  Interventions: Drug: quetiapine fumarate extended-release
- 2 (Experimental): quetiapine fumarate extended-release 300mg/Day1,600mg/Day2~6,administered once-daily
  Interventions: Drug: quetiapine fumarate extended-release
- 3 (Experimental): quetiapine fumarate extended-release 300mg/Day1,600mg/Day2,800mg/Day3~7,administered once-daily
  Interventions: Drug: quetiapine fumarate extended-release

INTERVENTIONS:
Drug: quetiapine fumarate extended-release — 200mg,oral,single dose
  Other Names: SEROQUEL XR
  Arms: 3
Drug: quetiapine fumarate extended-release — 300mg,oral,single dose
  Other Names: SEROQUEL XR

SUMMARY:
The primary objective of the study is to evaluate the pharmacokinetics of XR quetiapine fumarate(300mg,600mg,and 800mg once-daily) in Chinese schizophrenic patients .

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 through 60 years inclusive
* Schizophrenia diagnosis
* Body Mass Index (BMI) 20-27 kg/m2 (inclusive)
* Provision of written informed consent before initiation of any study

Exclusion Criteria:

* AIDS & hepatitis B
* History of seizure disorder
* History of episodic,idiopathic orthostatic hypotension

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2009-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
single dose PK parameters(300mg) | Day1 to 48 hour after Day 5
Steady-state multiple doses PK parameters | Day 1 to 48 hours after Day7

SECONDARY OUTCOMES:
Incidence and severity of AEs | sign ICF to Day 9
Clinical significant change in Lab test | baseline up to Day 9
Clinical significant change in vital signs | baseline up to Day 9

CONTACTS AND LOCATIONS:
Overall Officials: Tianmei Si, Principal Investigator — Peking University Institute of Mental Health
Locations (1):
- Research Site, Beijing, Beijing Municipality, China